CLINICAL TRIAL: NCT03858296
Title: Randomized Controlled Trial of Emotion Regulation for Inappropriate Anger Expression
Brief Title: Trial of Emotion Regulation for Inappropriate Anger Expression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Johan Bjureberg, Licenced Psychologist, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/2253-31/5
Record Dates: First submitted 2019-02-27; First posted 2019-02-28 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Inappropriate Anger Expression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Emotional awareness (Experimental): 4 modules of emotional awareness training
  Interventions: Behavioral: Internet-delivered emotional awareness training
- Cognitive reappraisal (Experimental): 4 modules cognitive reappraisal training
  Interventions: Behavioral: Internet-delivered Cognitive reappraisal training
- Awareness + reappraisal (Experimental): 4 modules emotional awareness and cognitive reappraisal training
  Interventions: Behavioral: Internet-delivered awareness and reappraisal training

INTERVENTIONS:
Behavioral: Internet-delivered emotional awareness training — Emotional awareness training is delivered via an internet platform during 4 weeks and includes therapist contact several times per week via the platform.
  Arms: Emotional awareness
Behavioral: Internet-delivered Cognitive reappraisal training — Cognitive reappraisal training is delivered via an internet platform during 4 weeks and includes therapist contact several times per week via the platform.
  Arms: Cognitive reappraisal
Behavioral: Internet-delivered awareness and reappraisal training — Emotional awareness and cognitive reappraisal training is delivered via an internet platform during 4 weeks and includes therapist contact several times per week via the platform.
  Arms: Awareness + reappraisal

SUMMARY:
The overall aim of the project is to develop three internet-delivered cognitive behavior therapies for inappropriate anger expression to test the isolated and combined effects of two types of regulation strategies, emotional awareness and cognitive reappraisal. Treatments will be evaluated in a stratified single blind parallel randomized block design, along with a pooled interrupted time series design. Self-recruited adults with elevated levels of anger will be stratified based on baseline level of anger. The particular aims are to examine:

1. the overall and separate effects of emotional awareness training, cognitive reappraisal training, and emotional awareness and cognitive reappraisal training on anger and aggression;
2. whether treatment effects are differentially moderated by baseline levels of emotional awareness, cognitive reappraisal, anger expression-out, anger expression-out, anger control-in, and trait anger;
3. whether the treatment effects are mediated by changes in emotional awareness, cognitive reappraisal, and anger control-in.

DETAILED DESCRIPTION:
1. Following the intention-to-treat principle, all primary data models will include all individuals as randomized. 3-month follow-up will be considered as the primary end-point. We will analyze both (1) overall treatment effect of all treatments (active treatment phase and 3-month follow-up compared to baseline) and (2) the relative efficacy for the emotional awareness training, cognitive reappraisal training, and emotional awareness and cognitive reappraisal training, respectively. We expect that, compared to a prolonged baseline phase, all treatments will result in greater improvements in on both primary and secondary outcomes. Further, we predict that the combined intervention will produce, on average, the strongest effects on primary and secondary outcomes relative to the separate interventions. We expect that cognitive reappraisal training will result in greater improvements relative to emotional awareness as a standalone treatment.
2. Growth models that include the interaction terms between experimental conditions (contrast coded) and baseline levels of moderator variables (as continuous measures) will be utilized to examine moderated treatment effects. Significant interactions will be examined following recommendations for probing interactions in growth models.
3. Weekly measurements of mediators will be analyzed with state-of-the-art methods for longitudinal mediation analysis, and we aim to to examine associations among process and outcome variables both within and between individuals as a function of condition and treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* experience of inappropriate anger expression that leads to significant distress or interferes with daily life (based on the STAXI-II)

Exclusion Criteria:

* risk for violent behavior that may harm others
* prior convictions of violence/abuse
* ongoing psychological treatment that may conflict with the offered treatment
* change in psychotropic medication within 2 months prior to enrollment
* severe psychiatric disorder, such as severe depression or risk of suicide
* alcohol or drug problems
* life circumstances that interfere with treatment (e.g., homeless)
* pronounced language skill deficits and learning difficulties (as the treatment format assumes normal reading and writing skills)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
State-Trait Anger Expression Inventory-2 (Subscales: Anger-out, Anger-in) | Change from baseline, once every week during treatment (0-4 weeks after baseline), and 3 months after treatment has ended.
  Levels of State-trait anger Expression. The subscales Anger Expression-Out (range: 8-32), Anger Expression-In (range: 8-32), and State Anger (range: 15-60) will be used, with higher scores indicating more anger.

SECONDARY OUTCOMES:
Emotion Regulation Questionnaire (Subscale: Reappraisal) | Change from baseline, once every week during treatment (0-4 weeks after baseline), and 3 months after treatment has ended.
  Levels of reappraisal from the subscale Reappraisal (range: 6-35, with higher scores indicating more reappraisal).
Five Facets Mindfulness Questionnaire (Subscales: Nonreactivity, Non-judging) | Change from baseline, once every week during treatment (0-4 weeks after baseline), and 3 months after treatment has ended.
  Levels of nonreactivity to inner experiences (range: 6-30; with higher scores indicating more nonreactivity) nonjudging of experience (range: 5-25; with higher scores indicating more nonjudging).
State-Trait Anger Expression Inventory-2 (Subscale: Anger control-in) | Change from baseline, once every week during treatment (0-4 weeks after baseline), and 3 months after treatment has ended.
  Levels of anger control-in (range: 8-32; higher scores indicating more anger control-in).
State-Trait Anger Expression Inventory-2 (Subscales: Trait anger, Anger control-out, State anger) | Change from baseline, 4 weeks after treatment starts, and 3 months after treatment has ended
  Levels of State-Trait Anger Expression. The subscales Trait Anger (range: 10-40; higher scores indicating more trait anger), Anger Control-Out (range: 8-32; higher scores indicating more anger control-out), State Anger (range: 15-60; higher scores indicating more anger control-in).
Aggression Questionnaire | Change from baseline, 4 weeks after treatment starts, and 3 months after treatment has ended. Ranges from 0-87, with higher higher scores indicating more aggression problems.
  Levels of aggression (range 0-87). Higher scores indicate more aggression.
Anger Rumination Scale | Change from baseline, 4 weeks after treatment starts, and 3 months after treatment has ended
  Levels of anger rumination (range: 19-76). Higher scores indicate more anger rumination.
Five Facets Mindfulness Questionnaire | Change from baseline, 4 weeks after treatment starts, and 3 months after treatment has ended
  Levels of mindfulness (range: 29-145). Higher scores indicate more mindfulness.
Emotion Regulation Questionnaire (Subscale Suppression) | Change from baseline, once every week during treatment (0-4 weeks after baseline), and 3 months after treatment has ended.
  Levels of suppression (range: 1-28). Higher scores indicate more suppression.
The Pittsburgh Sleep Quality Index | Change from baseline, 4 weeks after treatment starts, and 3 months after treatment has ended
  Sleep quality (range: 0-21). Higher scores indicate worse sleep quality.
Perceived Stress Scale 10 item version | Change from baseline, once every week during treatment (0-4 weeks after baseline), and 3 months after treatment has ended.
  Stress (range: 0-40). Higher scores indicate more negative stress.

OTHER OUTCOMES:
Treatment Credibility Scale | 1 week after treatment starts
  Treatment credibility and expectancy (range: 0-50) with higher scores indicating greater credibility/expectancy.
Client satisfaction Questionnaire | 4 weeks after treatment starts
  Levels of client treatment satisfaction (range: 8-32) with higher scores indicating more satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Bjureberg, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Centre for Psychiatry Research Karolinska Institutet and Stockholm County Council, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bjureberg J, Ojala O, Berg A, Edvardsson E, Kolbeinsson O, Molander O, Morin E, Nordgren L, Palme K, Sarnholm J, Wedin L, Ruck C, Gross JJ, Hesser H. Targeting maladaptive anger with brief therapist-supported internet-delivered emotion regulation treatments: A randomized controlled trial. J Consult Clin Psychol. 2023 May;91(5):254-266. doi: 10.1037/ccp0000769. Epub 2022 Nov 21. PMID 36409100